CLINICAL TRIAL: NCT06808841
Title: Sufentanil is Paired Via the BMP6/SMAD Pathway Cardiac Injury in Lower Extremity Fracture Surgery Function Study
Brief Title: Sufentanil in Patients With Lower Extremity Fracture Surgery Myocardial Damage Function Study
Acronym: Sipwlefsmdfs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, Professor, Second Hospital of Shanxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gz20250110
Record Dates: First submitted 2025-01-10; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Myocardial Injury
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low dose sufentanil group (Experimental): The concentration of sufentanil is set to concentration for the low-dose group
  Interventions: Drug: Sufentanil injection
- Medium-dose sufentanil group (Experimental): The concentration of sufentanil is set to medium-dose concentration for the low-dose group
  Interventions: Drug: Sufentanil injection
- High dose sufentanil group (Experimental): The concentration of sufentanil is set to high concentration for the low-dose group
  Interventions: Drug: Sufentanil injection
- Blank control group (Experimental): No analgesics were given
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sufentanil injection — Different concentrations of sufentanil were administered to three different subgroups of patients in the same way
  Other Names: Sufentanil dose
  Arms: High dose sufentanil group; Low dose sufentanil group; Medium-dose sufentanil group
Drug: Placebo — Placebo
  Arms: Blank control group

SUMMARY:
1. To analyze the association of different doses of opioids on myocardial injury/protection through BMP-6/SMAD pathway.
2. To observe the effect of different doses of opioids on the expression of BMP-6 in bone marrow.
3. To investigate the relationship between different doses of opioids and BMP-6 and perioperative cardiovascular adverse events in patients with lower extremity fracture surgery.

DETAILED DESCRIPTION:
This study explored the important role of BMP6/SMAD pathway in myocardial/injury protection by observing the effects of different doses of opioids on myocardial injury indexes hs-cTnI and BMP-6 related indexes in patients undergoing lower extremity fracture surgery, as well as the changes of BMP6 expression in bone marrow tissue of fracture end. The relationship between different doses of opioids and BMP6 and cardiac adverse events provides a theoretical basis for clinical rational drug use.

ELIGIBILITY:
Inclusion Criteria:

* There were 160 patients aged 18-65 years and older who needed surgery for lower extremity fracture.
* ASA grades I to III, gender is not limited.

Exclusion Criteria:

* Patients with acute myocardial infarction in the last 6 months, those with a history of heart failure, and those with elevated troponin levels before injury.
* Old fracture
* Stroke patients
* Liver cirrhosis, kidney failure
* Serious systemic infections, alcoholism, drug dependence
* Pathological fracture
* Use of glucocorticoids in the past one month
* Diabetic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-05 (Estimated); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Serum BMP6 | Immediate postoperative measurement
  Dose measurement of BMP6 in serum

SECONDARY OUTCOMES:
one marrow tissue BMP6 | Immediate postoperative measurement
  To observe the effect of different doses of opioids on the expression of BMP-6 in bone marrow tissue of fracture end

OTHER OUTCOMES:
Perioperative cardiac adverse events | Immediate postoperative measurement
  To observe the effects of opioids and BMP6 on perioperative cardiovascular adverse events (ACVE) in patients with lower extremity fractures

CONTACTS AND LOCATIONS:
Locations (1):
- Second Hospital of Shanxi Medical University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No